CLINICAL TRIAL: NCT05287334
Title: Measurement of Blood Loss Using Electrical Impedance Tomography
Brief Title: Blood Loss Measurement Using Electrical Impedance Tomography
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Czech Technical University in Prague (Other)
Collaborators: Military University Hospital, Prague (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 12229
Record Dates: First submitted 2022-03-10; First posted 2022-03-18 (Actual); Last update posted 2022-08-09 (Actual); Status verified 2022-08

CONDITIONS: Blood Loss
Keywords: Blood donation, EIT
MeSH Terms: conditions — Hemorrhage

STUDY DESIGN:
Intervention Model Description: Single group assignment. Approx 10-15 voluntary blood donors.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Voluntary blood donors (Experimental): Voluntary blood donors undergoing standard blood donation while measuring electrical impedance of the chest .
  Interventions: Device: Electrical impedance tomography measurement

INTERVENTIONS:
Device: Electrical impedance tomography measurement — During standard blood donation, donors' chest bioimpedance will be measured using electrical impedance tomography.

SUMMARY:
The project focuses on the possibility of detecting blood loss using electrical impedance tomography. Based on previous animal experiments, it was found that the bolus of saline significantly affects the signal of chest bioimpedance. It is assumed that blood loss of a similar volume will cause a similar signal change with the opposite trend. The aim of this project is to determine whether there is a significant change in the thoracic electrical impedance tomography signal when blood loss is caused by voluntary blood donation.

DETAILED DESCRIPTION:
Electrical impedance tomography is a bedside method of ventilation monitoring. The bioimpedance of the tissue depends, among other things, on its blood content. The area of the chest and especially the lungs is a heavily perfused tissue, which also serves as one of the reservoirs of blood in case of blood loss. It is therefore possible that blood loss will be visible on chest bioimpedance relatively soon.

The study will be performed on voluntary blood donors. Blood loss of 450 mL will be caused by the collection of donated blood. During blood collection at the transfusion department, thoracic bioimpedance will be measured using electrical impedance tomography. The resulting signal change will then be analyzed to determine the possibility of detecting and measuring blood loss using electrical impedance tomography.

ELIGIBILITY:
Inclusion Criteria:

* voluntary blood donation

Exclusion Criteria:

* standard exclusion criteria for voluntary blood donation based on the transfusion station protocol
* standard exclusion criteria for electrical impedance tomography according to the manufacturer

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2022-07-01 (Actual); Primary Completion 2022-10-10 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in chest electrical impedance due to blood loss. | Time frame of one voluntary blood donation process (15 min)
  A change in the electrical impedance of the chest of a voluntary blood donor caused by a blood donation.

CONTACTS AND LOCATIONS:
Overall Officials: Vaclav Ort, M.Eng., Principal Investigator — Czech Technical University in Prague, Fac. of Biomedical Engineering
Locations (2):
- Czechia (2):
  - Czech Technical University, Faculty of Biomedical Engineering, Kladno
  - Czech technical university in Prague, Facutly of biomedical engineering, Kladno

IPD SHARING:
Plan to Share IPD: No